CLINICAL TRIAL: NCT01044277
Title: Effect of Oral Glutathione Supplementation on the Levels of Blood Glutathione and Markers of Oxidative Stress in Healthy Adults (Glutathione Supplementation and Health (GSH) Study)
Brief Title: Oral Glutathione Supplementation on the Levels of Blood Glutathione
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, John P. Richie, Professor of Public Health Sciences and Pharmacology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PSHCI 09-059
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Healthy Adults
Keywords: glutathione; gluthathione peroxidases; GSH

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind - GSH 500 mg/GSH 125 mg/Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Glutathione supplementation-Double-Blind - GSH 500 mg/GSH 125 mg/Placebo
  Other name Gluthathione peroxidases
  Interventions: Drug: Glutathione supplementation
- Group B (Experimental): Glutathione supplementation-Double-Blind - GSH 500 mg/GSH 125 mg/Placebo
  Other name Gluthathione peroxidases
  Interventions: Drug: Gluthathione peroxidases
- Group C (Placebo Comparator): Placebo-Double-Blind - GSH 500 mg/GSH 125 mg/Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glutathione supplementation — 500 mg, two times daily
  Other Names: Gluthathione Peroxidates; GSH
  Arms: Group A
Drug: Gluthathione peroxidases — 125 mg, two times daily
  Other Names: Glutathione supplementation; GSH
  Arms: Group B
Other: Placebo — 2 times daily
  Other Names: Gluthathione peroxidases; GSH
  Arms: Group C

SUMMARY:
This trial is designed to provide evidence of the efficacy of glutathione supplementation and health(GSH) and includes the assessment of both short term and long term effects. Based on previous laboratory animal studies and clinical data, the investigators anticipate that the effects of oral GSH supplementation will be progressive and cumulative. The study will also allow for the evaluation of effects of withdrawal of the supplement on the outcome variables.

DETAILED DESCRIPTION:
This is a randomized double-blind, placebo-controlled study in which the treatment allocations will be kept sealed until the final statistical evaluation. The design will include the recruitment of 60 healthy subjects (30-79 yr of age) randomized into 3 groups. A total of 48 subjects, 16 per group will be required based upon power calculations and results from a previous clinical trial with selenium. An additional 4 subjects per group will be placed on trial to account for possible attrition or non-compliance. Blood, urine and exfoliated buccal mucosal samples will be obtained from all subjects at baseline. Questionnaire data on usual dietary intake will also be obtained at baseline. Eligible subjects will be required to have not have taken any high dose antioxidant supplements for at least 1 month prior to the study. Subjects will then begin supplementation according to the following schedule:

Group A, GSH (500 mg, 2 times daily); Group B, GSH (125 mg, 2 times daily); Group C, placebo (2 times daily). Eligible participants who sign the informed consent will be randomly assigned to either placebo or high or low dose Glutathione groups. Participants will be asked not to consume any other high-dose vitamin, multi-vitamin, or mineral supplements containing glutathione throughout the study in order to prevent variation in dose of supplemental GSH between subjects. Supplementation will continue for 6 months with biological samples collected at 1, 3 and 6 months after baseline. At 6 months, supplementation will be discontinued. A final collection of biological samples will occur 1 month afterwards. Compliance will be monitored by pill count.

Levels of glutathione will be measured in plasma, lymphocytes, and red blood cells as well as in exfoliated buccal mucosal cells. Biomarkers of oxidative stress will include blood levels of glutathionylated proteins and 8-isoprostanes and urine levels of 8-hydroxydeoxyguanosine. Glutamylcystine ligase and GST activities, and C-reactive protein will be determined in blood. Immune function biomarkers will be analyzed including t-natural killer cell cytotoxicity, lymphoproliferation, neutrophils phagocytosis, neutrophil respiratory burst assays.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and females between the ages of 30 and 79 years of age
* Not taking glutathione as a dietary supplement
* Not taking high dose antioxidant supplement prior to 1 month
* Baseline blood glutathione level of < 1 mmol/L

Exclusion Criteria:

* History or evidence of disease including cancer, diabetes, heart disease
* Subjects who smoke

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of glutathione on key biomarkers | 6 to 7 months
  Blood glutathione status

SECONDARY OUTCOMES:
Evaluations will be carried out to expand the above comparison by including adjustments for potential prognostic factors. | 6 to 7 months
  Biomarkers of oxidative stress and immune function

CONTACTS AND LOCATIONS:
Overall Officials: John P. Richie, Ph.D., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time we have no plan for sharing, however, if the need should arise, then sharing may be a possibility.

REFERENCES:
- [Derived] Richie JP Jr, Nichenametla S, Neidig W, Calcagnotto A, Haley JS, Schell TD, Muscat JE. Randomized controlled trial of oral glutathione supplementation on body stores of glutathione. Eur J Nutr. 2015 Mar;54(2):251-63. doi: 10.1007/s00394-014-0706-z. Epub 2014 May 5. PMID 24791752